CLINICAL TRIAL: NCT00290667
Title: 2-Weekly CHOP Chemotherapy With Dose-Dense Rituximab for the Treatment of Patients Aged 61 to 80 Years With Aggressive CD-20 Positive B-Cell Lymphomas: A Phase-II/Pharmacokinetic Study (CHOP-R-ESC)
Brief Title: Rituximab and Combination Chemotherapy in Treating Older Patients With Previously Untreated B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German High-Grade Non-Hodgkin's Lymphoma Study Group (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454505; DSHNHL-2004-1; EU-20536; DSHNHL-CHOP-R-ESC; EUDRACT-2005-00529-68
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage I adult Burkitt lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage IV adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Follicular | interventions — pegfilgrastim; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional: CHOP-14 + 8 x 2-weekly rituximab (Active Comparator): Arm I (2-weekly rituximab): Patients receive rituximab IV 375 mg/m^2 (females) and 500 mg/m^2 (males) over 4 hours on days 0, 14, 28, 42, 56, 70, 84, and 98. Patients also receive pegfilgrastim subcutaneously on day 4 of each course.
  Interventions: Biological: pegfilgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Other: pharmacological study; Radiation: radiation therapy
- Interventional: CHOP-14 + 8 x dose-dense rituximab (Active Comparator): Arm II (pharmacokinetic-based dose-dense rituximab): Patients receive rituximab IV 375 mg/m^2 (females) and 500 mg/m^2 (males) over 4 hours on days -1, 0, 3, 7, 14, 21, 28, and 42. Patients also receive pegfilgrastim subcutaneously on day 4 of each course.
  Interventions: Biological: pegfilgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Other: pharmacological study; Radiation: radiation therapy

INTERVENTIONS:
Biological: pegfilgrastim
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Other: pharmacological study
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, and prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with combination chemotherapy works in treating older patients with previously untreated B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine a pharmacokinetic profile for pharmacokinetics-based or rituximab within a CHOP-14 regimen comprising cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone in elderly patients with previously untreated aggressive B-cell lymphoma.
* To determine whether increased single-doses of rituximab for males can compensate their lower serum levels.
* Evaluate the safety and toxicity profile of this regimen in male patients.

Secondary

* Determine the rate of complete responses, primary progressions under therapy, event-free survival, progression-free survival, and overall survival in patients treated with this regimen.
* Determine the rate of primary progression in patients treated with this regimen.

OUTLINE: This is a multicenter study. All patients undergo the following treatment.

* Prephase treatment: Patients receive vincristine subcutaneously on day -6 and oral prednisone on days -6 to 0.
* Immunochemotherapy and radiotherapy: Patients receive CHOP chemotherapy comprising cyclophosphamide IV over 15 minutes, doxorubicin hydrochloride IV, and vincristine IV on day 1 and oral prednisone once daily on days 1-5. Patients also receive pegfilgrastim subcutaneously on days 4, 18, 32, 46, 60, and 74. Treatment with CHOP chemotherapy repeats every 14 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients who show no response after course 4 of CHOP chemotherapy proceed to salvage chemotherapy off study.

Patients are evaluated 2-4 weeks after completion of CHOP. Patients with initial bulky disease (i.e., diameter ≥ 7.5 cm) or extranodal involvement AND achieving complete remission (CR), unconfirmed CR (CRu), or partial remission undergo radiotherapy 5 days a week for 4 weeks. Patients who do not achieve CR or CRu 2 months after completion of radiotherapy proceed to salvage chemotherapy off study.

Patients are then stratified according to center, International Prognostic Index (1-2 vs 3-5), disease involvement (bulky vs extranodal vs bulky and/or extranodal), age (61-70 years old vs 71-80 years old), and gender. Patients are randomized to 1 of 2 treatment arms.

* Arm I (2-weekly rituximab): Patients receive rituximab IV 375 mg/m^2 (females) and 500 mg/m^2 (males) over 4 hours on days 0, 14, 28, 42, 56, 70, 84, and 98. Patients also receive pegfilgrastim subcutaneously on day 4 of each course.
* Arm II (pharmacokinetic-based dose-dense rituximab): Patients receive rituximab IV 375 mg/m^2 (females) and 500 mg/m^2 (males) over 4 hours on days -1, 0, 3, 7, 14, 21, 28, and 42. Patients also receive pegfilgrastim subcutaneously on day 4 of each course.

Some patients undergo blood sample collection periodically during and after treatment for pharmacokinetic studies.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then once a year therafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histological diagnosis of aggressive B-cell lymphoma

  * Previously untreated disease
  * Stage I-IV disease
* CD20-positive disease
* Any International Prognostic Index (IPI) score
* No secondary lymphoma after prior chemotherapy or radiotherapy
* No primary CNS lymphoma
* No primary gastrointestinal (MALT) lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* AST and ALT ≤ 3 times normal unless related to lymphoma
* Bilirubin ≤ 2 mg/dL unless related to lymphoma
* Creatinine ≤ 2 times normal unless related to lymphoma
* Fertile patients must use effective contraception
* No known allergic reactions against foreign proteins
* No active infections requiring systemically administered antibiotics or antiviral medications
* No noncompensated heart failure
* No dilatative cardiomyopathy
* No coronary heart disease with ST-segment depression in ECG
* No myocardial infarction during the past 6 months
* No chronic lung disease with hypoxemia
* No severe noncompensated hypertension
* No severe noncompensated diabetes mellitus
* No clinical signs of cerebral dysfunction
* No severe psychiatric disease
* No known HIV infection
* No active chronic hepatitis B or C infection
* No other concurrent diseases that exclude the administration of therapy as outlined by the study protocol

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 12 weeks since prior clinical trial participation
* No prior participation in this study
* No prior therapy, including murine antibody, for this cancer
* No prior organ transplantation
* No concurrent response-adapted radiotherapy ("iceberg radiotherapy")
* No other concurrent anticancer chemotherapy or other study medication

Ages: 61 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Actual)
Dates: Start 2004-02; Primary Completion 2013-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (in first 20 patients of each cohort with a distinct variation of the rituximab schedule) assessed on days -4, -1, 10, 29, 57, 99, 155, 239, 267, 295, 407, and 491 of treatment | -4 to 491 days of treatment
Safety and treatment related deaths at 3 months after study completion | 3 months after study completion
Toxicity assessed by NCI criteria, adverse events, serious adverse events, protocol adherence, and treatment-related deaths at 3 months after study completion | 3 months after study completion

SECONDARY OUTCOMES:
Time to treatment failure assessed at 2 years within the study and periodically thereafter | at 2 years within the study and periodically thereafterlif
Complete response rate assessed at 2 years within the study and periodically thereafter | at 2 years within the study and periodically thereafter
Progression rate | life-long
Survival time | life-long
Progression-free survival | life-long

CONTACTS AND LOCATIONS:
Overall Officials: Michael G.M. Pfreundschuh, MD, Study Chair — Universitaetsklinikum des Saarlandes; Norbert Schmitz, MD, PhD, Study Chair — Asklepios Klinik St. Georg
Locations (337):
- Czechia (2):
  - University Hospital Brno, Brno
  - Charles University Hospital, Prague
- Hopital Debrousse, Lyon, France
- Germany (323):
  - Haematologisch Onkologische Praxis, Aachen
  - Ostalb-Klinikum Aalen, Aalen
  - Klinikum St. Marien, Amberg
  - Gemeinschaftspraxis Fuer Innere Medizin, Haematologie Und Internistische Onkologie, Ansbach
  - Specialist Practice for Oncology, Aschaffenburg
  - II. Medizinische Klinik, Aschaffenburg
  - Haematologische Praxis, Augsburg
  - Hamatologische/Onkologische Gemeinschaftspraxis - Augsburg, Augsburg
  - Klinikum Augsburg, Augsburg
  - Kreiskrankenhaus Aurich, Aurich
  - Regional Hospital Bad Hersfeld, Bad Hersfeld
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - Internistische Praxis - Bad Salzuflen, Bad Salzuflen
  - Kreiskrankenhaus Bad Saeckingen, Bad Säckingen
  - Onkologische Schwerpunktpraxis und Tagesklinik Dres, Bad Soden
  - Ermstalklinik Bad Urach, Bad Urach
  - Klinikum am Bamberg, Bamberg
  - Krankenhaus Hohe Warte Mediziniche Klinik, Bayreuth
  - Klinikum Bayreuth, Bayreuth
  - Praxis Dr. med. Stefan Korsten, Bergisch Gladbach
  - Onkologisches Versorgungszentrum Friedrichshain, Berlin
  - DRK Kliniken Berlin - Koepenick, Berlin
  - Internistische Gemeinschaftspraxis - Berlin, Berlin
  - Haematologisch-Onkologische Schwerpunktpraxis, Berlin
  - Evang. Waldkrankenhaus Spandau, Berlin
  - Charite - Campus Charite Mitte, Berlin
  - Onkolog - Haematolog Schwerpunktpraxis, Berlin
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Vivantes Klinikum Neukoelln, Berlin
  - Robert Roessle Comprehensive Cancer Center - Charite Campus Buch, Berlin
  - Hospital Complex Bernburg, Bernburg
  - Franziskus Hospital, Bielefeld
  - Krankenhaus Bietigheim, Bietigheim
  - Saint Agnes Hospital, Bocholt
  - Augusta-Kranken-Anstalt gGmbH, Bochum
  - St. Josef-Hospital - Bochum, Bochum
  - Knappschaftskrankenhaus Bochum-Langendreer, Bochum
  - Johanniter-Krankenhaus Bonn, Bonn
  - Universitaetsklinikum Bonn, Bonn
  - Medizinische Poliklinik, Bonn
  - Praxis fuer Haematologie und Internistische Onkologie - Borken, Borken
  - Knappschaftskrankenhaus Bottrop, Bottrop
  - Hamatologische Sprechstunde, Brandenburg
  - Staedtisches Klinikum Braunschweig, Braunschweig
  - Praxis Dres. F.& G. Doering, Bremen
  - Klinikum Bremen-Mitte, Bremen
  - DIAKO Ev. Diakonie Krankenhaus gGmbH, Bremen
  - St. Joseph Hospital, Bremerhaven
  - Zentralkrankenhaus, Bremerhaven
  - Praxis fuer Haematologie und Onkologie - Burgwedel, Burgwedel
  - Medizinische Klinik am Lukas - Krankenhaus, Bünde
  - General Hospital, Celle
  - Onkologische Schwerpunktpraxis Celle, Celle
  - Hospital Kuchwald Chemnitz, Chemnitz
  - Klinikum Coburg, Coburg
  - Internistische Praxis - Coesfeld, Coesfeld
  - Praxis Internistischer Onkologie und Haematologie - Koeln, Cologne
  - Kliniken der Stadt Koeln gGmbH - Krankenhaus Holweide, Cologne
  - Praxis fuer Onkologie - Kalk, Cologne
  - Praxis Fuer Haematologie Internistische Onkologie, Cologne
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Lung Clinic Cologne-Merheim, Cologne-Merheim
  - Carl - Thiem - Klinkum Cottbus, Cottbus
  - Praxis Dr. Rheinhold Siegmund - Dr. Matthias Penke, Damme
  - Klinikum Darmstadt, Darmstadt
  - Staedtisches Klinikum Dessau, Dessau
  - Internistische Praxis, Detmold
  - Saint Johannes Hospital Dortmund, Dortmund
  - Klinikum Dortmund, Dortmund
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Johanniter-Krankenhaus Rheinhausen GmbH, Duisburg
  - St. Johannes Hospital - Medical Klinik II, Duisburg
  - Franz Hospital Dulmen, Dülmen
  - Florence-Nightingale-Krankenhause, Deaconess Kaiserswerth, Düsseldorf
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Klinikum Barnim GmbH, Werner Forssmann Krankenhaus, Eberswalde
  - Virngrund-Klinik Ellwangen, Ellwangen
  - Hans - Susemihl - Krankenhaus, Emden
  - Helios Klinikum Erfurt, Erfurt
  - Medizinische Klinik III - Universitaetsklinikum Erlangen, Erlangen
  - St. Antonius Hospital, Eschweiler
  - Universitaetsklinikum Essen, Essen
  - Evangelisches Krankenhaus Essen Werden, Essen
  - Staedtische Kliniken Esslingen, Esslingen am Neckar
  - Schwerpunktpraxis fuer Haematologie und Onkologie - Flensburg, Flensburg
  - Gemeinschaftspraxis fuer Internistische - Frankenthal, Frankenthal
  - Onkologie Bethanien, Frankfurt
  - Krankenhaus Nordwest, Frankfurt
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Klinikum Frankfurt (Oder) GmbH, Frankfurt (Oder)
  - St. Marienkrankenhaus - Frankfurt am Main, Frankfurt am Main
  - Praxis Internistischer Onkologie und Haematologie - Frechen, Frechen
  - Gemeinschaftspraxis - Freiburg, Freiburg im Breisgau
  - Evang. Deaconess Hospital Freiburg, Freiburg im Breisgau
  - Praxis fur Interdisziplinaere Onkologie, Freiburg im Breisgau
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Municipal Hospital Complex, Fulda
  - Klinikum Garmisch - Partenkirchen GmbH, Garmisch-Partenkirchen
  - Robert - Koch Hospital, Gehrden
  - Saint Josef Hospital, Gelsenkirchen
  - Internistische Praxisgemeinschaft, Germering
  - Centre for Internal Medicine Giessen, Giessen
  - Gemeinschaftspraxis Fuer Innere Medizin, Hematologie Und Onkologie, Giessen
  - Wilhelm-Anton-Hospital gGmbH, Goch, Goch
  - DR Herbert - Nieper Krankenhaus Goslar, Goslar
  - Staedtisches Klinikum Görlitz GmbH, Görlitz
  - Universitaetsklinikum Göttingen, Göttingen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Kreiskrankenhaus Gummersbach GMBH, Gummersbach
  - Internistisch-Haematologische Gemeinschaftspraxis - Gustrow, Güstrow
  - Staedtisches Klinikum Gütersloh, Gütersloh
  - Allgemeines Krankenhaus Hagen, Hagen
  - St. Marien Hospital - Katholisches Krankenhaus Hagen gGmbH, Hagen
  - St. Salvator Krankenhaus, Halberstadt
  - Internistische Gemeinschaftspraxis - Halle, Halle
  - Universitaetsklinikum Halle, Halle
  - Krankenhaus St. Elisabeth und St. Barbara, Halle
  - Krankenhaus Martha-Maria Halle-Doelau gGmbH, Halle
  - St. Sixtus Hospital, Haltern
  - Praxis fuer Innere Medizin - Bergedorf, Hamburg
  - Marienkrankenhaus, Hamburg
  - Allgemeines Krankenhaus Altona, Hamburg
  - Onkologische Schwerpunktpraxis Dr. med. Verpoort, PD Dr. med. Zeller and Dr. med. Wierecky, Hamburg
  - Asklepios Klinik St. Georg, Hamburg
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Asklepios Klinik Nord Heidberg, Hamburg
  - Haematologisch-Onkologische Praxis Altona, Hamburg
  - St. Marien Hospital, Hamm
  - Evangelische Krankenhaus Hamm, Hamm
  - Klinikum Stadt Hanau, Hanau
  - Schwerpunktpraxis Haematologie/Onkologie - Hannover, Hanover
  - Krankenhaus Siloah - Medizinische Klinik II, Hanover
  - Henriettenstiftung Frauenklinik, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Oncology Specialists Clinic, Harrislee
  - Ruprecht - Karls - Universitaet Heidelberg, Heidelberg
  - Thoraxklinik Heidelberg, Heidelberg
  - Regional Hospital Heidenheim, Heidenheim
  - Regional Hospital Am Plattenwald Bad Friedrichshall, Heilbronn
  - Klinikum Herford, Herford
  - Marienhospital at Ruhr University Bochum, Herne
  - Privatklinik Dr. R. Schindlbeck GmbH & Co. KG, Herrsching am Ammersee
  - Onkologische Schwerpunktpraxis, Hildesheim
  - St. Bernward Krankenhaus, Hildesheim
  - Staedtisches Krankenhaus Hildesheim, Hildesheim
  - Evang. Hospital, Holzminden
  - Haematologie und Internistische Onkologie Praxis, Homberg (Efze)
  - Universitaetsklinikum des Saarlandes, Homburg
  - Hospital Complex Hoyerswerda, Hoyerswerda
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Internistische Gemeinschaftspraxis - Jena, Jena
  - Klinikum der Friedrich-Schiller Universitaet Jena, Jena
  - Onkologische Gemeinschaftspraxis - Kaiserslautern, Kaiserslautern
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - St. Vincentius - Kliniken, Karlsruhe
  - Red Cross Hospital Kassel, Kassel
  - Internistische Gemeinschaftspraxis - Kassel, Kassel
  - Klinikum Kempten Oberallgaeu, Kempten
  - Staedtisches Krankenhaus Kiel, Kiel
  - Praxis fuer Haematologie und Onkologie, Koblenz
  - Stiftungsklinikum Mittelrhein - Gesundheitszentrum Evangelisches Stift Sankt Martin Koblenz gGmbH, Koblenz
  - Leonardis Clinic, Kornwestheim
  - Haematologische / Onkologische Schwerpunktpraxis, Krefeld
  - Klinikum Krefeld GmbH, Krefeld
  - Internistische Onkologische Praxis - Kronach, Kronach
  - Frankenwald Klinik, Kronach
  - Internistische Praxis - Landshut, Landshut
  - Klinikum Landshut, Landshut
  - Caritas - Krakenhaus Lebach, Lebach
  - Onkologische Schwerpunktpraxis - Leer, Leer
  - Praxis fuer Onkologie am Diakonissenhaus, Leipzig
  - Forschungsgesellschaft mbH, Leipzig
  - Gemeinschaftspraxis fuer Dres. Aldaoud und Schwarzer, Leipzig
  - University Leipzig Clinic of Internal Medicine, Leipzig
  - Klinikum "St. Georg" Leipzig, Leipzig
  - Klinikum Lippe - Lemgo, Lemgo
  - St. Vincenz Hospital Limburg, Limburg
  - St. Bonifatius Hospital Lingen, Lingen
  - Dreifaltigkeits Hospital, Lippstadt
  - Kreiskrankenhaus Loerrach, Loerrach
  - Onkologische Schwerpunktpraxis, Loerrach
  - Klinikum Ludwigsburg, Ludwigsburg
  - St. Marien Hospital Ludwighafen, Ludwigshafen
  - Klinikum der Stadt Ludwigshafen am Rhein, Ludwigshafen am Rhein
  - Schwerpunktpraxis fuer Haematologie und Onkologie - Luebeck, Lübeck
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Sana Kliniken Luebeck, Lübeck
  - Kreiskrankenhaus Luedenscheid, Lüdenscheid
  - Universitatsklinikum der MA, Magdeburg
  - Staedtisches Klinikum Magdeburg - Altstadt, Magdeburg
  - Internistische Gemeinschaftspraxis - Magdeburg, Magdeburg
  - St. Vincenz und Elisabeth Hospital, Mainz
  - Johannes Gutenberg University, Mainz
  - Gemeinschaftspraxis, Mannheim
  - III Medizinische Klinik Mannheim, Mannheim
  - Schwerpunktpraxis Internist Onkologie - Marburg, Marburg
  - Universitaetsklinikum Giessen und Marburg GmbH - Marburg, Marburg
  - Regional Hospital Mayen, Mayen
  - Gemeinschaftspraxis Dres. med. Ellbrueck/Goeller/Kraenzle/Niedermeier/Jocham, Memmingen
  - Krankenhaus Ludmillenstift, Meppen
  - Gemeinschaftspraxis - Minden, Minden
  - Klinikum Minden, Minden
  - Ev. Hospital Bethesda, Mönchengladbach
  - Krankenhaus Maria Hilf GmbH, Mönchengladbach
  - Haematologische Praxis - Moenchengladbach, Mönchengladbach
  - Universitaets - Kinderpoliklinik, Munich
  - Krankenhaus Muenchen Schwabing, Munich
  - Munich Oncologic Practice at Elisenhof, Munich
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Staedtisches Krankenhaus Muenchen - Harlaching, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Municipal Hospital Munich, Munich
  - Klinikum Schwaebisch Gmuend Stauferklinik, Mutlangen
  - Evangelisches Krankenhaus - Muelheim, Mülheim
  - St. Marien Hospital - Muelheim an der Ruhr, Mülheim
  - Kreiskrankenhaus Muenchberg, Münchberg
  - Gemeinschaftspraxis - Muenster, Münster
  - Haematologisch - Onkologische Gemeinschaftspraxis - Muenster, Münster
  - Klinik und Poliklinik fuer Kinder und Jugendmedizin - Universitaetsklinikum Muenster, Münster
  - Staedtisches Krankenhaus Nettetal GmbH, Nettetal
  - Klinikum Neubrandenburg, Neubrandenburg
  - Onkologische Schwerwpunktpraxis Dr. Ladda, Neumarkt
  - Regional Hospital Neumarkt, Neumarkt
  - Onkologische Schwerpunktpraxis Dr. Schmidt, Neunkirchen
  - Staedtisches Klinikum Neunkirchen gGmbH, Neunkirchen
  - Internistische Praxis - Neuss, Neuss
  - Lukaskrankenhaus Neuss, Neuss
  - DRK Krankenhaus Neuwied, Neuwied
  - Praxis fuer Haematologie und Interne Onkologie, Norderstedt
  - Gemeinschaftspraxis fuer Onkologie - Nordhorn, Nordhorn
  - Gemeinschaftspraxis fuer Haematologie - Northeim, Northeim
  - Praxisklinik fuer Innere Medizin - Nuernberg, Nuremberg
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Schlossbergkliniken Oberstaufen, Oberstaufen
  - Internistische Gemeinschaftspraxis - Offenbach, Offenbach
  - Klinikum Offenburg, Offenburg
  - Pius Hospital - Oldenburg, Oldenburg
  - Internistische Gemeinschaftspraxis - Oldenburg, Oldenburg
  - Ev. Hospital Oldenburg, Oldenburg
  - Klinikum Oldenburg, Oldenburg
  - St. Martinus Hospital - Olpe, Olpe
  - Marien Hospital, Osnabrück
  - Klinikum Osnabrück GmbH, Osnabrück
  - Paracelsus - Klinik Osnabrück, Osnabrück
  - Bruederkrankenhaus St. Josef Paderborn, Paderborn
  - Asklepios Klinik - Parchim, Parchim
  - Staedtisches Krankenhaus, Pforzheim
  - Krankenhaus Siloah - Pforzheim, Pforzheim
  - Praxis fuer Innere Medizin am Krankenhaus Siloah - Pforzheim, Pforzheim
  - Gemeinschaftspraxis - Pinneberg, Pinneberg
  - Klinikum Ernst Von Bergmann, Potsdam
  - Kreiskrankenhaus Radebeul, Radebeul
  - Gemeinschaftspraxis - Ravensburg, Ravensburg
  - Krankenhaus St. Elisabeth - Ravensburg, Ravensburg
  - Elisabeth Krankenhaus, Recklinghausen
  - Prosper-Hospital Recklinghausen, Recklinghausen
  - Hematologische Onkologische Praxis, Regensburg
  - Klinikum der Universitaet Regensburg, Regensburg
  - Krankenhaus Barmherzige Brueder Regensburg, Regensburg
  - Internistische Praxis Dres. Hempel und Hochdorfer, Rehling
  - Klinikum Remscheid GmbH, Remscheid
  - Jakobi Krankenhaus, Rheine
  - Haematologische/Onkologische Schwerpunktpraxis - Rostock, Rostock
  - Klinik und Poliklinik fuer Innere Medizin - Universitaet Rostock, Rostock
  - Klinikum Suedstadt Rostock, Rostock
  - Diakonie - Krankenhaus, Rotenburg (Wümme)
  - Internistische Schwerpunktpraxis, Rüsselsheim am Main
  - Gemeinschaftspraxis - Saarbruecken, Saarbrücken
  - Caritasklinik St. Theresia, Saarbrücken
  - St. Elizabeth-Klinik Saarlouis, Saarlouis
  - Martin - Luther Hospital, Schleswig
  - Praxis fur Innere Medizin - Schmiedeberg, Schmiedeberg
  - Deaconess Hospital, Schwäbisch Hall
  - Gemeinschaftspraxis fuer Haematologie und Internist - Schweinfurt, Schweinfurt
  - Leopoldina - Krankenhaus, Schweinfurt
  - HELIOS Klinikum - Schwelm, Schwelm
  - Klinikum Schwerin, Schwerin
  - St. Marien - Krankenhaus Siegen GMBH, Siegen
  - Evang. Jung-Stilling Hospital, Siegen
  - St. Lukas - Clinic Solingen, Solingen
  - Krankenhaus Maria-Hilf - Stadtlohn, Stadtlohn
  - Onkologische Schwerpunktpraxis - Straubing, Straubing
  - Hospital Bad Cannstatt, Stuttgart
  - Haematologische Praxis, Stuttgart
  - Klinik fuer Onkologie - Katharinenhospital Stuttgart, Stuttgart
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Gastroenterologische und Haematologisch-Onkologische Praxis E. M. Dr. Hoering von Ehr Respondek, Stuttgart
  - Klinikum Stuttgart - Buergerhospital, Stuttgart
  - Robert-Bosch-Krankenhaus, Stuttgart
  - St. Elisabeth Hospital Thuine, Thuine
  - Regional Hospital Traunstein, Traunstein
  - Onkologische Gemeinschaftspraxis - Trier, Trier
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Krankenhaus Der Barmherzigen Brueder, Trier
  - Praxis Fuer Internistische Haematologie / Onkologie, Troisdorf
  - Hospital Tutzing, Tutzing
  - Universitaetsklinikum Tuebingen, Tübingen
  - Praxis fuer Haematologie und Onkologie, Twistringen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Ev. Hospital Unna, Unna
  - St. Marienhospital - Vechta, Vechta
  - Onkologische Schwerpunktpraxis - Villingen, Villingen
  - Municipal Hospital Complex, Villingen-Schwenningen
  - Regional Hospital Waldbrol, Waldbröl
  - Haematologische Praxis, Weiden
  - Gemeinschaftspraxis feur Haemotologie und Onkologie - Weilheim, Weilheim
  - Sophien - und Hufeland - Klinikum Weimar gGmbH, Weimar
  - Onkologische Schwerpunktpraxis, Wendlingen
  - Harz-Klinikum Wernigerode-Blankenburg GmbH, Wernigerode
  - Asklepios Nordseeklinik Westerland GmbH, Westerland
  - Ammerland-Klinik GmbH, Westerstede
  - Hospital Wetzler, Wetzlar
  - Deutsche Klinik fuer Diagnostik, Wiesbaden
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
  - Ev. Hospital Witten-Herdecke, Witten
  - Evangelisches Krankenhaus - Lutherstadt Wittenberg, Wittenberg
  - Klinikum der Stadt Wolfsburg, Wolfsburg
  - Burkhard and Reimann Gemeinschaftspraxis, Worms
  - Helios Kliniken Wuppertal University Hospital, Wuppertal
  - Kliniken St. Antonius, Wuppertal
  - Medizinische Poliklinik, Universitaet Wuerzburg, Würzburg
  - Heinrich-Braun-Krankenhaus Zwickau, Zwickau
- Azienda Ospedaliera di Padova, Padua, Italy
- Erasmus MC - Sophia Children's Hospital, Rotterdam, Netherlands
- Akademia Medyczna im. Piastow Slaskich, Wroclaw, Poland
- Goeteborg University, Gothenburg, Sweden
- Switzerland (6):
  - Kantonsspital Aarau, Aarau
  - Universitaets-Kinderspital beider Basel, Basel
  - Ospedale "la Carita", Locarno, Locarno
  - Kinderspital Luzern, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - University Children's Hospital, Zurich
- Royal Manchester Children's Hospital, Manchester, England, United Kingdom